CLINICAL TRIAL: NCT03326284
Title: Optimizing Per Meal Protein Intake During Weight Loss
Brief Title: Optimal Protein Dose Per Meal During Weight Loss in Perspective to Maintaining Muscle Mass
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: Arla Foods (Industry); Innovation foundation (Unknown); Mejeribrugets ForskningsFond (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 57403
Record Dates: First submitted 2017-05-08; First posted 2017-10-31 (Actual); Last update posted 2019-07-31 (Actual); Status verified 2018-06

CONDITIONS: Protein Metabolism
Keywords: Hypocaloric diet; Dietary protein

STUDY DESIGN:
Intervention Model Description: : Forty women (~ 50 years) will be randomized to four groups. Following a five day hypocaloric diet (three groups) or an energy balanced diet (one group). The women will report to the laboratory to ingest one of three different protein doses.
Who Masked: Participant
Masking Description: The protein doses provided will be masked. As all participants will receive the same amount and the drinks will taste similarly.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- 15g protein hypocaloric diet (Experimental): Following a 5-day hypocaloric diet the subjects (n=10) will ingest 15g of protein and their mixed muscle protein synthesis response will be monitored using tracer kinetics.
  Interventions: Other: 15 g protein hypocaloric
- 35g protein hypocaloric diet (Experimental): Following a 5-day hypocaloric diet the subjects (n=10) will ingest 35g of protein and their mixed muscle protein synthesis response will be monitored using tracer kinetics.
  Interventions: Other: 35 g protein hypocaloric
- 60g protein hypocaloric diet (Experimental): Following a 5-day hypocaloric diet the subjects (n=10) will ingest 60g of protein and their mixed muscle protein synthesis response will be monitored using tracer kinetics.
  Interventions: Other: 60 g protein hypocaloric
- 35g protein energy balanced diet (Experimental): Following a 5-day energy balanced diet the subjects (n=10) will ingest 35g of protein and their mixed muscle protein synthesis response will be monitored using tracer kinetics.
  Interventions: Other: 35 g protein energy balance

INTERVENTIONS:
Other: 15 g protein hypocaloric — Following a 5 day hypocaloric diet one group of 10 women will ingest 15 g of protein
  Arms: 15g protein hypocaloric diet
Other: 35 g protein hypocaloric — Following a 5 day hypocaloric diet one group of 10 women will ingest 35 g of protein
  Arms: 35g protein hypocaloric diet
Other: 60 g protein hypocaloric — Following a 5 day hypocaloric diet one group of 10 women will ingest 60 g of protein
  Arms: 60g protein hypocaloric diet
Other: 35 g protein energy balance — Following a 5 day energy balanced diet one group of 10 women will ingest 35 g of protein
  Arms: 35g protein energy balanced diet

SUMMARY:
The primary aim of the trial is to determine the optimal dose of protein per meal in relation to enhancing muscle protein synthesis and thereby in perspective counteract muscle loss during weight loss. In addition, we aim to determine whether the response to protein intake is reduced in women on hypocaloric diet compared to in women on an energy-balanced diet.

DETAILED DESCRIPTION:
Aim of this project is to determine the optimal protein dose (high quality milk protein) per meal in relation to enhancing muscle protein synthesis and thereby counteract muscle loss during weight loss.

The hypothesis is that the optimum dose of protein for women on a hypocaloric diet will be greater than when women eat an energy sufficient diet, and also higher than the optimal dose previously determined in weight stable men.

Methods: Forty women (~ 50 years) will be randomized to four groups. Following a five day hypocaloric diet (three groups) or an energy balanced diet (one group). The women will report to the laboratory to ingest one of three different protein doses. The muscle protein response to the different doses of protein will be determined by the muscle protein fractional synthetic rates using tracer kinetics.

ELIGIBILITY:
Inclusion Criteria:

* healthy
* Postmenopausal women

Exclusion Criteria:

* Smoking
* Metabolic and/or chronic diseases

Ages: 45 Years to 75 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2018-02-01 (Actual); Study Completion 2018-02-01 (Actual)

PRIMARY OUTCOMES:
Fractional synthetic rate | 3 hours after ingestion of protein
  Mixed muscle protein synthetic rate determined by tracer kinetics

SECONDARY OUTCOMES:
Muscle signalling | 3 hours after ingestion of protein.
  Markers for myofibrillar protein turnover measured by RT-PCR and western blotting

CONTACTS AND LOCATIONS:
Locations (1):
- Aarhus University, Department for Public Health, Section for Sport Science, Aarhus, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Larsen MS, Witard OC, Holm L, Scaife P, Hansen R, Smith K, Tipton KD, Mose M, Bengtsen MB, Lauritsen KM, Mikkelsen UR, Hansen M. Dose-Response of Myofibrillar Protein Synthesis To Ingested Whey Protein During Energy Restriction in Overweight Postmenopausal Women: A Randomized, Controlled Trial. J Nutr. 2023 Nov;153(11):3173-3184. doi: 10.1016/j.tjnut.2023.08.011. Epub 2023 Aug 19. PMID 37598750